CLINICAL TRIAL: NCT01557712
Title: Estimate the Efficiency of the Association of an Injection of Ketamine and the Venlafaxine in the Severe Major Depressive Disorder for Six Weeks.
Acronym: KETADEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1129
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine+venlafaxine (Experimental): one injection of 0.5 mg/kg of kentamine the first day plus venlafaxine (150-375 mg day) during 6 weeks
  Interventions: Drug: ketamine venlafaxine
- venlafaxine (Active Comparator): venlafaxine (150-375 mg day) during 6 weeks
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: ketamine venlafaxine — After a washout period of 7 days of psychotropic medications with the exception of cyamemazine and hydroxyzine:
  * Intravenous injection on day 0 to 0.5 mg / kg of ketamine
  * D0 to D4: 75 mg of venlafaxine
  * D4 to D14: 150 mg per day of venlafaxine
  * D14 to D42: 150 mg daily of venlafaxine to 375 mg per day of venlafaxine if patient not responder
  Arms: Ketamine+venlafaxine
Drug: Venlafaxine — After a washout period of 7 days of psychotropic medications with the exception of cyamemazine and hydroxyzine:
  * Intravenous injection on day 0 to 0.5 mg / kg of placebo (saline serum)
  * D0 to D4: 75 mg of venlafaxine
  * D4 to D14: 150 mg per day of venlafaxine
  * D14 to D42: 150 mg daily of venlafaxine to 375 mg per day of venlafaxine if patient not responder
  Arms: venlafaxine

SUMMARY:
The objective of this study is to evaluate the effectiveness of ketamine (infusion of 0.5mg/kg) and venlafaxine compared to the use of venlafaxine alone in the treatment of major depression (MADRS score ≥ 20 ) to six weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over,
* Introducing a single depressive episode or recurrent unipolar
* Responding to the diagnosis of severe major depressive episode according to DSM IV (Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition): MADRS score ≥ 20,
* absence of treatment with ketamine for analgesia or anesthesia during the last 6 months
* Affiliate (or beneficiary) to a social security system
* Informed consent signed

Exclusion Criteria:

* Contraindication to ketamine administration or treatment with venlafaxine;
* Failure of treatment with venlafaxine in the current episode (as low as 150 mg for 15 days);
* Axis I diagnosis according to DSM IV bipolar disorder (type I, II or III), schizoaffective disorder, schizophrenia, alcohol and other toxic or weaned for at least 6 months;
* Current Episode resistant stage V according to the classification of Thase and Rush (failed a course of bilateral ECT);
* Major depressive episode with severity criteria (significant risk of suicide is a MADRS score ≥ 5-SI; decubitus complications, intravenous hydration);
* episode currently being treated with fluoxetine;
* Patients hospitalized without their consent or measure of legal protection (guardianship, curatorship);
* Affection Organic likely to affect cognitive abilities and brain structures (eg, HIV, MS, lupus, Parkinson's disease, epilepsy, dementia ...) or decompensation;
* Pregnancy or breastfeeding underway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Depressive state | 6 weeks
  Assessment of depression by MADRS defining six weeks:
  * the state of clinical response defined by a MADRS score less than 50% in MADRS score at baseline initial set.
  * the state of clinical remission is defined by obtaining a MADRS score ≤ 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire, Grenoble, France